CLINICAL TRIAL: NCT00710879
Title: A Study to Evaluate the Clinical Performance of a Multi-Purpose Solution.
Brief Title: Evaluation of a Multi-Purpose Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 568
Record Dates: First submitted 2008-06-30; First posted 2008-07-08 (Estimated); Results first posted 2011-02-08 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Contact Lens Solutions
Keywords: Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multipurpose Solution (Experimental): Multi-purpose solution administered to adapted FDA group I soft contact lens wearers and FDA group IV soft contact lens wearers.
  Interventions: Device: Bausch & Lomb Multi-Purpose Solution

INTERVENTIONS:
Device: Bausch & Lomb Multi-Purpose Solution — Daily care for contact lenses.

SUMMARY:
This study evaluates a multi-purpose solution when used on a daily wear basis by currently adapted soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Is an adapted Group I or Group IV soft contact lens wearer and agrees to wear the study lenses on a daily wear basis.
* Must be able and willing to comply with all treatment and follow-up study procedures.
* Must have a clear central cornea.
* VA correctable to 0.3 LogMar or better (driving vision)

Exclusion Criteria:

* Systemic disease affecting ocular health.
* Using systemic or topical medications.
* Wear monovision, multifocal or toric contact lenses.
* Any grade 2 or greater slit lamp findings.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bev Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Dr. Nicholas Marsico, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled in this study on 07/07/2008 and last subject exited on 02/02/2009. 180 participants were enrolled at 9 investigative sites in the United States.
Pre-assignment Details: This study focused on participants of Japanese descent (at least one grandparent born in Japan) for a minimum of 20% of total enrollment. 180 participants were enrolled, 3 participants were ineligible at screening, 177 participants were eligible at the start of the study.
Groups:
- Multi-purpose Solution and Optima 38 Lenses: Multi-purpose solution when used on a daily wear basis with United States (US) Food and Drug Administration (FDA) Group I contact lenses (Optima 38) with no scheduled replacement. Participants were followed for 3 months.
- Multi-Purpose Solution and Acuvue 2 Lenses: B&L Multi-Purpose Solution when used on a daily wear basis with United States (US) Food and Drug Administration (FDA) Group IV contact lenses (Acuvue 2) with scheduled replacements every 2 weeks. Participants were followed for 6 months.
Period: Overall Study
Arm/Group | Multi-purpose Solution and Optima 38 Lenses | Multi-Purpose Solution and Acuvue 2 Lenses
Started | 60 | 117
Completed | 58 | 113
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multi-purpose Solution and Optima 38 Lenses | Multi-Purpose Solution and Acuvue 2 Lenses | Total
Number analyzed (Participants) | 60 | 117 | 177
Age, Customized [Number; unit: Participants]
  Aged 18-64 | 60 (11.0) | 117 (10.3) | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 75 | 112
  Male | 23 | 42 | 65
Participants with Grandparents Born in Japan [Number; unit: Participants] — Participants with Grandparents Born in Japan
  Participants
    1 Grandparent | 0 | 11 | 11
    2 Grandparents | 7 | 18 | 25
    3 Grandparents | 4 | 6 | 10
    4 Grandparents | 49 | 82 | 131

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Efficacy
Description: Excellent = No bacterial infection suspected and no ocular pathogens detected and bacteria of normal flora <0-103 CFU/mL. Good = No bacterial infection suspected and no ocular pathogens detected and bacteria of normal flora <103-105 CFU/mL. Skeptical = Bacterial infection suspected and ocular pathogens detected and bacteria of normal flora ≥ 105 CFU/mL. No Efficacy = Bacterial infection definite and ocular pathogens detected and bacteria of normal flora ≥ 105 CFU/mL. Pathogens were H. aegyptius, H. influenzae, Moraxella spp., P. aeruginosa, S. pneumoniae, S. aureus, N. gonorrhoeae
Time Frame: 2 weeks, 3 months
Population: All eligible, dispensed eyes with cultures taken within window. Group I subjects were cultured at the 3-Month Visit. Group IV subjects were cultured at the 2-week Follow-up visit.
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | Multi-purpose Solution and Optima 38 Lenses | Multi-Purpose Solution and Acuvue 2 Lenses
Number analyzed (Participants) | 58 | 113
Number analyzed (eyes) | 115 | 226
Eyes
  Excellent | 114 | 219
  Good | 0 | 3
  Skeptical | 1 | 4
  No Efficacy | 0 | 0

2. Secondary Outcome: Solution Related AE's and Lens Changes
Description: Very Safe = No solution related AEs and no changes in lens properties related to the solution. Safe = No solution related AEs and slight change in lens properties related to the solution, but lens wear was continued. Skeptical = Solution related AEs were suspected and lens properties changed due to the solution and lens wear was discontinued. Not Safe = Solution related AEs were present and lens properties changed due to the solution and lens wear was discontinued.
Time Frame: 3 months, 6 months
Population: All Eligible, Dispensed Eyes
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | Multi-purpose Solution and Optima 38 Lenses | Multi-Purpose Solution and Acuvue 2 Lenses
Number analyzed (Participants) | 60 | 120
Number analyzed (eyes) | 120 | 240
Eyes
  Very Safe | 118 | 238
  Safe | 2 | 2
  Skeptical | 0 | 0
  Not Safe | 0 | 0

3. Secondary Outcome: Solution Utlility
Description: The Utility was determined based on the results of the efficacy and safety evaluations.
Time Frame: 3 months, 6 months
Population: All Eligible, Dispensed Eyes
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Multi-purpose Solution and Optima 38 Lenses | Multi-Purpose Solution and Acuvue 2 Lenses
Number analyzed (Participants) | 58 | 117
Number analyzed (Eyes) | 115 | 234
Eyes
  Very Useful | 112 | 225
  Useful | 2 | 5
  Slightly Useful | 1 | 4
  Not Useful | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated at every visit. Group 1, 3 months and group 4, 6 months.
Arm/Group | Multi-purpose Solution and Optima 38 Lenses | Multi-Purpose Solution and Acuvue 2 Lenses
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/240
Other Adverse Events (participants affected / at risk) | 0/120 | 0/240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.